CLINICAL TRIAL: NCT01040962
Title: Fall Risk Assessment in People With Diabetic Neuropathy
Status: Completed | Type: Observational
Sponsor: Stephen D. Jernigan, PT, PhD (Other)
Responsible Party: Sponsor-Investigator, Stephen D. Jernigan, PT, PhD, Clinical Assistant Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Other Study IDs: 11481; GCRC Protocol #0122 (Other: University of Kansas Medical Center)
Record Dates: First submitted 2009-12-28; First posted 2009-12-30 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: neuropathy; diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Falls Risk Assessment, Diabetic Peripheral Neuropathy Patients

SUMMARY:
Fall risk is increased in people with diabetic peripheral neuropathy (DPN) and yet, minimal research has been conducted to identify appropriate fall risk assessment tools and improve our understanding of falls in these individuals. Purpose: The primary purpose of this study is to establish a foundation of knowledge needed to address falls in people with DPN. This will be accomplished through 1) comparing the validity of 4 fall risk assessment tools, 2) identifying risk factors for falls and 3) determining how quality of life is influenced by factors related to falls in people with DPN.

DETAILED DESCRIPTION:
All subjects participate in testing that involves questionnaires, cognitive testing, fall risk assessment, and other testing related to physical parameters including body mass index, glycosylated hemoglobin, lower extremity nerve conduction study, and ankle range of motion, proprioception and strength. After testing, subjects are interviewed to determine fall status (faller or non-faller). A "faller" is defined as someone that has fallen at least 2 times in the past year. Data Analysis: The validity of the fall risk assessment tools will be compared using sensitivity and specificity analyses. Variables related to ankle function, neuropathy, glycemic control and general activity will be analyzed for association with recent fall history through multivariable logistic regression. Variables related to falls, neuropathy and activity level will be analyzed for association with health-related quality of life through multivariable linear regression.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with diabetic peripheral neuropathy

Exclusion Criteria:

* major medical depression
* non-diabetes related musculoskeletal problems that limit ambulation
* open wounds on the weight bearing surfaces of the feet
* requires another person's assistance to walk
* uncorrected visual deficits that influence gait and/or balance
* history of stroke or other CNS pathology that impairs gait and/or balance
* diagnosed untreated vestibular disorder that results in gait and/or balance disturbances

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons that have diabetic peripheral neuropathy
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2008-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Jernigan, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - North Kansas City Hospital, Kansas City, Missouri